CLINICAL TRIAL: NCT06179329
Title: No-Touch Saphenous Venous Harvesting TechniQue versUs Radial artEry in Coronary Artery Bypass Grafting in womEN: The QUEEN Multicenter Randomized Controlled Trial
Brief Title: One-year Patency Comparison Between Radial Artery and No-touch Saphenous Vein Grafts in Women Undergoing Isolated CABG
Acronym: QUEEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto Nacional de Cardiologia (Unknown); Hospital Unimed João Pessoa (Unknown); Hospital do Coração Alagoano Prof. Adib Jatene (Unknown); Hospital Hernan Henriquez Aravena (Unknown); Hospital Norte Paranaense (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5723/23/125
Record Dates: First submitted 2023-12-06; First posted 2023-12-21 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Disease; Surgery-Complications; Graft Failure
Keywords: Cardiovascular Surgery; Coronary Disease; Women; Graft patency
MeSH Terms: conditions — Heart Diseases; Coronary Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial - Anterolateral / Saphenous - RCA (Other): Radial artery graft for the anterolateral wall, and "no-touch" saphenous vein graft for the right coronary artery territory
  Interventions: Procedure: Coronary artery bypass graft
- Radial - RCA / Saphenous - Anterolateral (Other): Radial artery graft for the territory of the right coronary artery and "no-touch" saphenous vein for the anterolateral wall.
  Interventions: Procedure: Coronary artery bypass graft

INTERVENTIONS:
Procedure: Coronary artery bypass graft — Randomization will be performed for stratification according to the target coronary arteries and the randomly determined block size from 4 to 6. The randomization result will be delivered in a sealed envelope in the operating room (before the time out) for one of the two drawn strategies.

SUMMARY:
The use of a graft from the left internal thoracic artery to the left anterior descending artery has become the gold standard for the indication of coronary artery bypass grafting. However, choosing a graft for the second-best coronary artery, focusing on long-term patency, is still a challenge. The saphenous vein using the "no-touch" technique is an alternative to a radial artery graft, but there is little evidence, especially in women. This randomized clinical study aims to compare the patency of these grafts in the second-best coronary artery in women undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18 years or older and younger than 75 years, undergoing isolated and primary myocardial revascularization surgery, with triarterial coronary artery disease (three vessels involved) in vessels subject to surgical revascularization and left ventricular ejection fraction greater than 35%. The target coronary vessels of the study will be those in the territory of the left circumflex artery and the right coronary artery, which must have at least 1.5 mm in diameter, and with proximal obstructive lesions of at least 70%.

Exclusion Criteria:

1. Preoperative conditions:

   1. Lack of the patient's written informed consent.
   2. Presence of poorly controlled diabetes, with a glycated hemoglobin value >8 mg/dl.
   3. Emergency or salvage surgery, where the intervention needs to be performed quickly due to the critical clinical condition of the patient.
   4. Renal failure with glomerular filtration rate (creatinine clearance) <30 mL/min.
2. Inability to use the saphenous and/or radial vein

   1. Positive Allen test using a pulse oximeter
   2. Presence of abnormal flow detected by means of a Doppler exam in one of the grafts to be used.
   3. History of vasculitis or Raynaud's syndrome, varicose veins, or history of previous saphenous vein removal
3. Conditions that may affect patient follow-up

   1. Presence of advanced peripheral arterial disease
   2. Known contrast allergy: Presence of a documented allergy to the contrast agent used in radiological procedures.
   3. Impossibility of tracking due to geographic inaccessibility.
   4. Patients with lack of adherence to guidelines and/or prescribed medications.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
One Follow-up with angiography | One year after surgery
  The primary endpoint will be the proportion of saphenous vein and radial artery grafts that were completely occluded on follow-up angiography

SECONDARY OUTCOMES:
Evaluate in-hospital clinical outcomes 30 days after CABG | Thirty days after surgery
  Death from any cause, perioperative myocardial infarction (occurring between 0 and 30 days), late myocardial infarction (occurring between 31 days and 1 year), reoperation of surgical revascularization and/or coronary angioplasty.
  Hand claudication and thenar paresthesia, complications potentially related to radial artery extraction, will be reported according to the specific diagnoses and confirmed with a consulting neurologist. As all patients will receive a radial artery graft, clinical events will be reported for the entire study population.

CONTACTS AND LOCATIONS:
Overall Officials: Omar AV Mejia, MD, PhD, Principal Investigator — InCor - Instituto do Coração do Hospital das Clínicas da FMUSP
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No